CLINICAL TRIAL: NCT03501485
Title: Impact of Protein Supplementation to Mother Milk on Resting Energy Expenditure (REE) in Growing Healthy Preterm Infants.
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Tel-Aviv Sourasky Medical Center (Other Government)
Responsible Party: Sponsor
Other Study IDs: 0741-16-TLV-DM
Record Dates: First submitted 2018-02-06; First posted 2018-04-18 (Actual); Last update posted 2020-06-16 (Actual); Status verified 2019-07

CONDITIONS: Infant,Premature
MeSH Terms: conditions — Premature Birth

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Resting Energy Expenditure is the amount of energy, usually expressed in Kcal required for a 24 hour period by the body during resting conditions. It is closely related to, but not identical to, basal metabolic rate.

According to the ESPGHAN committee guidelines on enteral nutrient supply for preterm infants, which were published in 2010, the daily protein intake of extremely low birth weight infants shall be 4.5 g/kg/day, and for those above 1000g, 4 g/kg/day. In order to meet these recommendations, the human milk for all premature infants is enriched with human milk fortifier, and supplemental liquid protein according to our NICU protocol.

Little is known on the effect of this enrichment on the basal metabolic rate of premature infants.

One way of determining the basal metabolic rate is by measuring the resting energy expenditure. In order to do that the investigators use an indirect calorimety by using the Deltatrac II metabolic monitor (Datex-Ohmeda). This instrument uses the principle of the open-circuit system that allows continuous measurements of oxygen consumption and carbon dioxide production using a constant flow generator.

DETAILED DESCRIPTION:
Infants will be enrolled when tolerating full feeds (150-160 ml/kg/d) of human breast milk fortified with standard fortifier for 2 days and before protein supplementation.

Metabolic studies will be conducted while the infants are prone and asleep and at the same time of the day (noon time) for all infants, starting 1 hour after the completion of the last feed. Measurements will be stopped during body movements.

Each measure, once a day, will last for 30 min. A total of 4 REE measurements will be performed for all participants: before starting with protein supplementation, on day 0 (D0), and at days 2, 3 and 4 of protein supplementation.

ELIGIBILITY:
Inclusion Criteria:

* Preterm infants born with birth weight < 1500 g gestation
* Full enteral feeds (150-160 ml/kg/d) of breast milk fortified with standard HM fortifier will be well tolerated for 2 days, without significantly gastric residuals (less than 5%)
* Clinically and thermally stable.

Exclusion Criteria:

* Ventilated infant (invasive or non-invasive)
* Necrotizing enterocolitis (NEC)
* IVH grade 3-4
* BPD
* PDA
* Active infection.
* Congenital or genetic disorder ( trisomy, heart defect.)

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Healthy, appropriate weight for gestational age, gavage-fed, preterm infants
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2017-12-18 (Actual); Primary Completion 2022-01-01 (Estimated); Study Completion 2022-02-01 (Estimated)

PRIMARY OUTCOMES:
Changes in metabolic measurements | At day 0, 2, 3, 4
  Changes in metabolic measurements through indirect calorimetry using using a Deltatrac II metabolic monitor from baseline at day 0, throughout day 2, 3 and 4.

CONTACTS AND LOCATIONS:
Overall Officials: Dror Mandel, MD, Principal Investigator — Tel-Aviv Sourasky Medical Center
Locations (1):
- Department of Neonatology Tel Aviv Medical Center, Tel Aviv, Israel